CLINICAL TRIAL: NCT01895764
Title: Effect of the Combination of Methotrexate and Adalimumab on Reduction of Immunization in Ankylosing Spondylitis (COMARIS)
Acronym: COMARIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRI12-ED-COMARIS; 2012-004939-23 (EudraCT Number); A130042-32 (Other: ANSM); 2012-R41 (Other: CPP)
Record Dates: First submitted 2013-04-24; First posted 2013-07-10 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab (Active Comparator): adalimumab 40mg every 2 weeks
  Interventions: Drug: Adalimumab
- Adalimumab + Methotrexate (Experimental): adalimumab 40mg every 2 weeks and methotrexate 10mg per week
  Interventions: Drug: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Adalimumab — adalimumab, subcutaneous injection, 40mg every 2 weeks, week 0 until week 26
  Other Names: Humira
Drug: Methotrexate — methotrexate, subcutaneous injection, 10mg per week, week -2 until week 26
  Other Names: Metoject
  Arms: Adalimumab + Methotrexate

SUMMARY:
The purpose of this study is to determine if association of methotrexate with adalimumab leads to decrease immunogenicity beside adalimumab alone in Ankylosing Spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age or older
* Able and willing to give written informed consent and to comply with the requirements of the study protocol
* Subject met the definition of Ankylosing Spondylitis (AS) based on ASAS Criteria
* Subject with active AS, has had an inadequate response, an intolerance or an to one or more nonsteroidal anti-inflammatory drugs

Exclusion Criteria:

* Previous adalimumab treatment or previous treatment with more than one anti TNF alpha therapy.
* Previous methotrexate treatment, not stopped 3 month before inclusion
* Surgery scheduled during study
* Female subject without method of contraception
* Contraindication to adalimumab or methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-04-27 (Actual)

PRIMARY OUTCOMES:
presence or absence of antibodies against adalimumab | 6 months

SECONDARY OUTCOMES:
Change from baseline of the Ankylosing Spondylitis Disease Activity Score (ASDAS) | 6 months
Change from baseline of T and B cells concentrations. | 6 months
Change from baseline of "APRIL" and "TNF alpha" concentrations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilie DUCOURAU, MD, Principal Investigator — CHRU de TOURS
Locations (11):
- France (11):
  - Rhumatologie, CH de BLOIS, Blois
  - Rhumatologie, CHRU de BREST, Brest
  - Rhumatologie, CHD LA ROCHE SUR YON, La Roche-sur-Yon
  - Rhumatologie, CHR du MANS, Le Mans
  - Rhumatologie, CHRU de NANTES, Nantes
  - Rhumatologie / IPROS, CHR d'ORLEANS, Orléans
  - Rhumatologie, CHRU de POITIERS, Poitiers
  - Rhumatologie, CHRU de RENNES, Rennes
  - Rhumatologie, CH de SAINT BRIEUC, Saint-Brieuc
  - Médecine polyvalente, CH de SAINT NAZAIRE, Saint-Nazaire
  - Rhumatologie, CHRU de TOURS, Tours

REFERENCES:
- [Result] Ducourau E, Rispens T, Samain M, Dernis E, Le Guilchard F, Andras L, Perdriger A, Lespessailles E, Martin A, Cormier G, Armingeat T, Devauchelle-Pensec V, Gervais E, Le Goff B, de Vries A, Piver E, Paintaud G, Desvignes C, Ternant D, Watier H, Goupille P, Mulleman D. Methotrexate effect on immunogenicity and long-term maintenance of adalimumab in axial spondyloarthritis: a multicentric randomised trial. RMD Open. 2020 Jan;6(1):e001047. doi: 10.1136/rmdopen-2019-001047. Epub 2020 Jan 9. PMID 31958280